CLINICAL TRIAL: NCT03642158
Title: Targeted Transcranial Magnetic Stimulation for Cognitive Rehabilitation After Traumatic Brain Injury
Brief Title: rTMS for Cognitive Rehabilitation After TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Virginia Commonwealth Neurotrauma Initiative (Unknown)
Responsible Party: Principal Investigator, George Gitchel, Director of Clinical Research, Parksinon's Disease Education, Research and Clinical Center (PADRECC), Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 02332
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Cognitive Impairment; Traumatic Brain Injury
MeSH Terms: conditions — Cognitive Dysfunction; Brain Injuries, Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active TMS (Active Comparator): Subjects receive rTMS over the right DLPFC, in 2 second bursts at 10 Hz, followed by a 19 second break, for a total of 20 minutes. Stimulator intensity is set to 80% of motor threshold on day one, and 100% of motor threshold for the remainder of intervention. This paradigm is continued for 5 consecutive days.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation
- Sham TMS (Sham Comparator): Identical to active arm, but stimulator intensity is reduced to 30% of motor threshold, and the stimulator coil is oriented tangentially to the skull to "stimulate" air space above the head instead of cortical tissue.
  Interventions: Device: repetitive Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: repetitive Transcranial Magnetic Stimulation — repetitive Transcranial Magnetic Stimulation (rTMS) utilizes a magnetic coil of wire to non-invasively and painlessly activate small sections of the brain through the skull.

SUMMARY:
A novel and promising therapy for cognitive dysfunction is non-invasive brain stimulation, of which transcranial magnetic stimulation (TMS) is a form. TMS is currently FDA-approved for use in depression and migraine. It is under investigation for use in a number of other neurologic and psychiatric disorders. In addition to its potential to improve affective symptoms, recent research has suggested that TMS targeted to select cortical regions can also improve cognition. In trials of TMS therapy for psychiatric disorders, several studies have shown benefits for cognitive function alongside symptom amelioration. In healthy persons, a course of stimulation of the parietal area improved objective measures of learning and memory. Among persons with TBI, there have been case reports supporting improvement in cognitive function and postconcussive symptoms; however, there have not yet been any controlled studies of TMS for TBI-related cognitive dysfunction.

DETAILED DESCRIPTION:
Subjects with a history of TBI will be recruited into this double-blind, sham controlled, crossover with washout study design. Study will involve one week (5 consecutive days) of treatment, a 7 day off period, followed by a second week of rTMS treatment. Motor threshold will determine level of stimulation, and active rTMS stimulation will occur of the right DLPFC. Subjects will be paid for their time.

ELIGIBILITY:
Inclusion Criteria:

1. one or more mild to moderate TBIs*;
2. at least one year but no more than 20 years from worst injury;
3. ability to complete cognitive and neurophysiological testing;
4. available for duration of study;
5. between 18 and 65 years of age;
6. mild or greater cognitive symptoms on the TBI-QOL Cognition General Concerns scale

Exclusion Criteria:

1. severe or penetrating TBI;
2. history of psychotic or manic illness;
3. history of intracranial surgery;
4. history of skull fracture;
5. history of seizures in candidate or candidate's family
6. ferrous metallic implants or implantable medical device;
7. medications that are known to reduce seizure threshold;
8. pregnancy.
9. history of multiple sclerosis, stroke, brain tumor, epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Auditory target detection task | 10 minutes
  subjects listen to a series of sounds, and will monitor for a specific sounds.
Ruffs 2 and 7 selective attention test | ~5 minutes
  subjects must visually search for the numbers 2 and 7 among other distractors.
DKEFS Verbal Fluency | 10 minutes
  a measure of internal search and selection process, requires subject to generate several lists of items.
California Verbal Learning Test II | 10 minutes
  subjects are required to learn and recall an unfamiliar word list.

SECONDARY OUTCOMES:
EEG | 10 minutes
  resting state power spectra of EEG will be collected to analyze.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Holmes McGuire Veterans Affairs Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No